CLINICAL TRIAL: NCT04452760
Title: Effects of Ten-Weeks Progressive Resistance Training on Neuromuscular Performance, Mobility, Heart Rate Variability and Sleep Quality in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jacobo Á. Rubio, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCAM-CE071923
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis
Keywords: neurological disorders; resistance training; strength training; sleep quality; neuromuscular performance; functional capacity
MeSH Terms: conditions — Multiple Sclerosis; Nervous System Diseases; Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Only testing sessions
  Interventions: Other: Testing sessions
- Progressive resistance training group (Experimental): 10-weeks of progressive resistance training group. Leg press, leg extension, calf raises, hip extension exercises.
  Interventions: Other: Physical exercise; Other: Testing sessions

INTERVENTIONS:
Other: Physical exercise — Physical exercise intervention
  Arms: Progressive resistance training group
Other: Testing sessions — Testing sessions

SUMMARY:
Multiple Sclerosis (ME) is a degenerative, inflammatory and autoimmune demyelinating disease of the central nervous system, characterized by demyelination due to inflammation and degeneration of the myelin sheaths enveloping nerves of the eye, periventricular grey matter, brain, spinal cord and brainstem. The symptoms associated with MS include symptomatic fatigue, muscle weakness, ataxia, mobility and balance problems or cognitive problems. Strength training has been shown to improve strength and mobility in persons with MS.

DETAILED DESCRIPTION:
Multiple Sclerosis (ME) is a degenerative, inflammatory and autoimmune demyelinating disease of the central nervous system, characterized by demyelination due to inflammation and degeneration of the myelin sheaths enveloping nerves of the eye, periventricular grey matter, brain, spinal cord and brainstem. The symptoms associated with MS include symptomatic fatigue, muscle weakness, ataxia, mobility and balance problems or cognitive problems. Resistance training has been shown to improve strength, sleep quality and mobility in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* mild or moderate disability with clinical mild spastic-ataxic gait disorder.
* stable phase of the disease.

Exclusion Criteria:

* Expanded Disability Status Scale (EDSS) < 6.
* relapsing disease within the preceding 12 months.
* corticosteroid treatment within the last months before study inclusion.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction of Knee Extension | Before the program training
  the maximum force (N) that can be produced voluntarily by the knee extension muscles during an isometric contraction is measured. The leg of the participant is fixed to an isokinetic device, and the participant makes a 5-second attempt, developing all the strength he or she can.
Maximal Voluntary Isometric Contraction of Knee Extension | After 10 weeks
  the maximum force (N) that can be produced voluntarily by the knee extension muscles during an isometric contraction is measured. The leg of the participant is fixed to an isokinetic device, and the participant makes a 5-second attempt, developing all the strength he or she can.
Rate of Force Development | Before the program training
  Rate of force development in knee extension
Rate of Force Development | After 10 weeks
  Rate of force development in knee extension
Central Activation Ratio | Before the program training
  The central activation ratio (CAR) was determined using superimposed electrical stimulation during maximum voluntary contractions
Central Activation Ratio | After 10 weeks
  The central activation ratio (CAR) was determined using superimposed electrical stimulation during maximum voluntary contractions
Spasticity | Before the program training
  Pendulum test
Spasticity | After 10 weeks
  Pendulum test

SECONDARY OUTCOMES:
Walking speed | Before the program training
  Test 10 m-walks
Walking speed | After 10 weeks
  Test 10 m-walks
Static Balance | Before the program training
  Romberg Test with eyes open and closed. Analysis with force plates
Static Balance | After 10 weeks
  Romberg Test with eyes open and closed. Analysis with force plates
Functional capacity | Before the program training
  Sit-to-Stand Test
Functional capacity | After 10 weeks
  Sit-to-Stand Test
Heart Rate Variability | Before the program training
  Sleeping Heart Rate Variability
Heart Rate Variability | After 10 weeks
  Sleeping Heart Rate Variability
Sleep Quality | Before the program training
  Acelerometry and Karolinska Sleep Diary
Sleep Quality | After 10 weeks
  Acelerometry and Karolinska Sleep Diary

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Á Rubio-Arias, Dr, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data will be published in a journal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the completion of study
Access Criteria: The data will be published in a journal

REFERENCES:
- [Derived] Andreu-Caravaca L, Ramos-Campo DJ, Chung LH, Rubio-Arias JA. Can strength training modify voluntary activation, contractile properties and spasticity in Multiple Sclerosis?: A randomized controlled trial. Physiol Behav. 2022 Oct 15;255:113932. doi: 10.1016/j.physbeh.2022.113932. Epub 2022 Jul 27. PMID 35905806
- [Derived] Andreu-Caravaca L, Ramos-Campo DJ, Abellan-Aynes O, Avila-Gandia V, Chung LH, Manonelles P, Rubio-Arias JA. 10-Weeks of resistance training improves sleep quality and cardiac autonomic control in persons with multiple sclerosis. Disabil Rehabil. 2022 Sep;44(18):5241-5249. doi: 10.1080/09638288.2021.1934738. Epub 2021 Jun 9. PMID 34107841